CLINICAL TRIAL: NCT03602027
Title: Dose Climbing Trial of Anlotinib Plus Gefitinib in the First-line Treatment of Advanced Gene Positive Non-squamous Non-small Cell Lung Cancer
Brief Title: Phase I Study of the Combination of Anlotinib With Gefitinib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTERL007
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — anlotinib; Gefitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Plus Gefitinib (Experimental): This study will include a sequential evaluation of 3 subjects per dose group. low-dose groups: Anlotinib 8mg per day and Gefitinib. middle-dose groups: Anlotinib 10mg per day and Gefitinib. high-dose groups: Anlotinib 12mg per day and Gefitinib.
  A dose limiting toxicity (DLT) event is defined as any of the following events:
  1. CTCAE Grade 4 event (ANC<1000/ul, body temperature≥38.5°C);
  2. Grade 3 non-hematologic toxicity (except for nausea and vomiting that could be improved with optimal supportive care, escalation of alkaline phosphatase) If a DLT is experienced in any dose group, the cohort will be expanded to 6 subjects. If 2 DLTs are experienced in any dose group, the dose escalation ceased. The MTD was defined as the dose having at most two out of six patients experience DLT.
  Interventions: Drug: Anlotinib; Drug: Gefitinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 8mg p.o. qd in low-dose groups (3 subjects). 10mg p.o. qd in middle-dose groups (3 subjects). 12mg p.o. qd in high-dose groups (3 subjects).
Drug: Gefitinib — Gefitinib 250mg orally daily for three weeks

SUMMARY:
The purpose of this clinical study is to evaluate the tolerability and toxicity of different dose of Anlotinib puls Gefitinib in First-line Treatment of Advanced Gene Positive Non-squamous Non-small Cell Lung Cancer , to provide a reference of dosage for Phase II clinical trials

DETAILED DESCRIPTION:
This is a randomized, single -center study conducted in China to compare the tolerability and toxicity of different dose of Anlotinib Plus Gefitinib in patients of Advanced GenePositive Non-squamous Non-small Cell Lung Cancer.From low dose group up to high dose group, each one had 3 patients at least.Primary group received anlotinib 8mg. The dose of Anlotinib would increase gradually until MTD. Eligible patients were instructed to take Gefitinib 250mg orally daily for three weeks and 8mg/10mg/12mg Anlotinib orally daily on day 1 to 14 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Be≥18 years of age on the day of signing informed consent and With good compliance and agree to accept follow-up of disease progression and adverse events.
* Patients with histologic or cytologic confirmation of advanced or metastatic NSCLC with stage III or IV disease.（For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment）
* Epidermal Growth Factor Receptor(EGFR)mutations confirmed by molecular detection (including, but not limited to, 20 exon, 19 exon deletion and L858R) external pathological examination was accepted (including pathological or blood test results)
* Patients have not been received systematic treatment，including chemotherapy and EGFR -TKIs（Tyrosine kinase inhibitors）
* There were at least one target lesions in the past three months has not yet accepted radiotherapy, and could be recorded by magnetic resonance imaging (MRI) or computer tomography (CT) measuring accurately at least in one direction(The maximum diameter needs to be recorded), including conventional CT ≥20 mm or spiral CT ≥10 mm.
* Life expectancy ≥3 months.
* Have a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* With normal marrow, liver ,renal and coagulation function:
* The blood routine examination need to be standard (no blood transfusion and blood products within 14 days, no g-csf and other hematopoietic stimulating factor correction)
* Hemoglobin（HB）≥90 g/L
* A Neutrophil count of （ANC）≥1.5×109/L
* A Platelet count of （PLT）≥80×109/L
* A Total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL)
* A alanine aminotransferase (ALAT) and a aspartate aminotransferase (ASAT) of ≤2.5 UNL, in case of liver metastasis ALAT and ASAT≤5 UNL
* A creatinine (Cr) of ≤1.5 UNL; a creatinine clearance rate ≥ 60ml/min (Cockcroft-Gault)
* Doppler echocardiography: left ventricular ejection fraction (LVEF) is lower than normal (50%)
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.

Exclusion Criteria:

* Small cell lung cancer (include Small cell lung cancer mixture of NSCLC).
* Iconography (CT or MRI) shows that the tumor vessels have 5 mm or less, or Cardiovascular involvement by Central tumor ; Or obvious lung empty or necrotic tumor.
* Patients has a history of malignant tumors. Patients with basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma, or cervical cancer in situ who have undergone possible curative treatment and have not suffered any recurrence of the disease within 5 years from the start of treatment.
* Patients with Other active malignant tumors requiring concurrent treatment
* Patients who have not recovered to grade 1 or below after previous systemic antitumor therapy (except alopecia)
* Patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (14 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage)
* Uncontrollable hypertensive (systolic blood pressure or greater 140 mmHg or diastolic blood pressure or greater 90 mmHg, despite the best drug treatment)
* Significant cardiac disease as defined as: grade II or greater myocardial infarction, unstable arrhythmia(Including corrected QT interval (QTc )period between male or greater 450 ms, female or greater 470 ms); New York Heart Association (NYHA) grade II or greater heart dysfunction , or Echocardiography reveal left ventricular ejection fraction （LVEF）Less than 50%
* Patients with grade II or greater peripheral neuropathy, except due to trauma
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) >Upper Limit of Normal( ULN)+ 4 seconds or APTT（activated partial thromboplastin time ） ULN > 1.5, with bleeding tendency or be treated with thrombolysis and anticoagulation.

Note: under the premise of International Normalized ratio (INR) of prothrombin time (PT) Less than or equal to 1.5, allow to administrate low-dose heparin (adult daily dose is 06000 ~ 12000 U) or low-dose aspirin (100 mg daily dosage or less) , for prophylactic purposes

* Urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours
* Patients with respiratory syndrome (difficulty breathing of level 2 or higher ), serous cavity effusion need to surgical treatment ( including pleural of level 2 or higher with respiratory distress and anoxia, need for intubation or pleurodesis treatment, severe ascites of level 2 need to surgery invasive treatment, pericardial of level 2 and affect physiological function)
* Patients with severe infections , and need to receive systemic antibiotic treatment.（ the infection with grade 2 or above and requiring intravenous antibacterial therapy ）;Decompensated diabetes or other contraindication with high dose glucocorticoid therapy）
* Active or chronic hepatitis c and/or Hepatitis B virus (HBV) infection
* Serious, non-healing wound, ulcer, or bone fracture
* Has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* Has received major surgery or severe traumatic injury, fractures or ulcer Within 4weeks before Random
* Patients have participated in other antitumor drug clinical trials Within 4 weeks before enrollment or prepare to receive systemic anti-tumor treatment during the study or Within 4 weeks before randomization, including cytotoxic therapy cellular, Signal transduction inhibitors, immune therapy (or receiving mitomycin C Within six weeks before taking experimental drug therapy).Field overspread radiotherapy (ef-rt) was carried out within 4 weeks before the grouping or limited field radiotherapy was carried out within 2 weeks before the grouping to evaluate tumor lesions
* Severe weight loss (> 10%) Within 6 weeks before Random
* Has Clinically significant hemoptysis Within 3 months before Random (daily hemoptysis than 50 ml;Or significant clinical significance of bleeding symptoms or have definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, baseline period + + and above of fecal occult blood, or vasculitis, etc.
* Has venous thromboembolism events Within 12 months before Random, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* Patients who have a history of mental drug abuse and cannot be cured or have mental disorders
* There are any contraindications with receiving anlotinib or gefitinib treatment
* There are allergic reaction to contrast media, anlotinib, and/or excipient of experimental drug
* There are allergic reaction to the contrast agent
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | From enrollment to completion of study. Estimated about 4 months.
  Dose Limiting Toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria
Maximum tolerance dose | From enrollment to completion of study. Estimated about 4 months
  Maximum Tolerance Dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DLT reported.

SECONDARY OUTCOMES:
disease control rate | From enrollment to 2 months after treatment
  Clinical response of treatment according to RESIST v1.1 criteria (DCR, disease control rate)
time to progression | From enrollment to progression of disease. Estimated about 6 months
  The length of time from enrollment until the time of progression of disease (TTP, time to progression).